CLINICAL TRIAL: NCT07282509
Title: A Phase Ib/II Clinical Trial to Evaluate the Safety and Efficacy of Transcatheter Arterial Infusion of Paclitaxel Cationic Liposome Combined With Systemic Therapy in Participants With Advanced Hepatocellular Carcinoma for Second-line Treatment
Brief Title: Safety and Efficacy of Paclitaxel Liposome Arterial Infusion Combined With Systemic Therapy for Second-Line Treatment of Advanced Liver Cancer
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HA131-005
Record Dates: First submitted 2025-11-21; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Advanced Hepatocellular Carcinoma (HCC)
MeSH Terms: interventions — pembrolizumab; lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Phase Ib Cohort 1 (Experimental): Lenvatinib combined with elonstobart.
  Interventions: Drug: Enlonstobart Injection; Drug: Lenvatinib Mesilate Capsules
- Phase Ib Cohort 2 (Experimental): Transcatheter arterial infusion of HA131 combined with systemic therapy (lenvatinib with pembrolizumab).
  Interventions: Drug: HA131; Drug: Pembrolizumab Injection; Drug: Lenvatinib Mesilate Capsules
- Phase Ib Cohort 3 (Experimental): Transcatheter arterial infusion of HA131 combined with systemic therapy (lenvatinib with elonstobart )
  Interventions: Drug: HA131; Drug: Enlonstobart Injection; Drug: Lenvatinib Mesilate Capsules
- Phase II Experimental Arm (Experimental): Transcatheter arterial infusion of HA131 combined with systemic therapy (lenvatinib with or without elonstobart ).
  Interventions: Drug: HA131; Drug: Enlonstobart Injection; Drug: Lenvatinib Mesilate Capsules
- Phase II Control Arm (Active Comparator): Systemic therapy alone (lenvatinib with or without elonstobart ).
  Interventions: Drug: Enlonstobart Injection; Drug: Lenvatinib Mesilate Capsules

INTERVENTIONS:
Drug: HA131 — Phase Ib: Dose escalation. Phase II: Administration at the RP2D dose determined in Phase Ib. Transcatheter Arterial Infusion.
  Arms: Phase II Experimental Arm; Phase Ib Cohort 2; Phase Ib Cohort 3
Drug: Enlonstobart Injection — Administered via intravenous infusion.
  Arms: Phase II Control Arm; Phase II Experimental Arm; Phase Ib Cohort 1; Phase Ib Cohort 3
Drug: Pembrolizumab Injection — Administered via intravenous infusion.
  Arms: Phase Ib Cohort 2
Drug: Lenvatinib Mesilate Capsules — Administered orally.

SUMMARY:
This trial is an open-label, dose-escalation, and randomized controlled Phase Ib/II clinical study for second-line treatment in participants with advanced hepatocellular carcinoma (HCC). Its primary objective is to evaluate the safety, tolerability, pharmacokinetic profiles, and efficacy of transcatheter arterial infusion of HA131 combined with systemic therapy in the second-line treatment of participants with advanced HCC.

ELIGIBILITY:
Inclusion Criteria:

* 1.Aged 18 to 75 years (inclusive), regardless of gender;
* 2.Diagnosed with hepatocellular carcinoma (HCC) by histopathology, cytology, or imaging;
* 3.HCC classified as B/C stage per BCLC (Barcelona Clinic Liver Cancer) staging system, or IIb/IIIa/IIIb stage as defined in Clinical Practice Guidelines for Primary Liver Cancer (2024 Edition) (organized by the Guidelines Committee of the Chinese Society of Clinical Oncology, 2024);
* 4.Child-Pugh liver function class ≤ 7 points within 7 days prior to the first dose administration;
* 5.Progressive disease after prior first-line systemic antineoplastic therapy containing PD-1/PD-L1 monoclonal antibody;
* 6.At least one measurable lesion at the hepatic arterial infusion site per RECIST (Response Evaluation Criteria in Solid Tumors) Version 1.1 (lesion longest diameter ≥ 1 cm; lesions that have not received prior local therapy, or lesions that progressed again after local therapy);
* 7.ECOG (Eastern Cooperative Oncology Group) Performance Status (PS) score: 0-1.
* 8.Controlled hypertension, with blood pressure ≤ 150/90 mmHg and no changes to the antihypertensive regimen within one week prior to screening;
* 9.Estimated survival time of more than 3 months;
* 10.Before randomization, major organ/system functions are basically normal, meeting the criteria as assessed by laboratory tests.
* 11.Eligible individuals of childbearing potential (both males and females) must agree to use reliable contraceptive methods (hormonal contraceptives, barrier methods, or abstinence) with their partners during the trial and for at least 6 months after the last dose; female individuals of childbearing age must have a negative serum pregnancy test within 7 days before enrollment;
* 12.Participants must be informed about the study prior to the trial and voluntarily sign a written informed consent form.

Exclusion Criteria:

* 1.Pathologically confirmed fibrolamellar hepatocellular carcinoma (HCC), sarcomatoid HCC, cholangiocellular carcinoma, or combined hepatocellular-cholangiocarcinoma;
* 2.History of liver surgery and/or local treatment for HCC within 4 weeks prior to the first dose;
* 3.Previous antineoplastic treatment with lenvatinib;
* 4.Use of traditional Chinese medicine (TCM) preparations with indicated efficacy for anti-HCC within 14 days prior to the first dose; having received immune checkpoint inhibitors within 28 days prior to the first dose.
* 5.Active brain metastases, leptomeningeal disease, or uncontrolled spinal cord compression;
* 6.Adverse reactions from previous antineoplastic treatment that have not resolved to ≤ Grade 1 per NCI-CTCAE Version 5.0 (except for toxicities such as alopecia that are deemed to pose no safety risks by the investigator);
* 7.Contraindications to transcatheter arterial infusion interventional surgery; known contraindications or severe allergic reactions to any component of lenvatinib, PD-1/PD-L1 monoclonal antibody, paclitaxel, or cationic liposomes;
* 8.Malabsorption syndrome or inability to take oral medications due to other reasons;
* 9.Need for administration of strong inducers or strong inhibitors of CYP2C8 and CYP3A4 within 2 weeks prior to the first study treatment or during the treatment period;
* 10.Active infection within 2 weeks prior to the first dose; presence of peripheral neuropathy of Grade II or higher (per NCI-CTCAE Version 5.0);
* 11.History of autoimmune disease, immunodeficiency, other acquired or congenital immunodeficiency diseases, or current use of immunosuppressants;
* 12.Untreated active hepatitis B.
* 13.Participants positive for anti-hepatitis C virus antibody (HCV-Ab) with HCV-RNA level above the lower limit of the central laboratory's detection range;
* 14.Participants with active syphilis;
* 15.A history of past or current hepatic encephalopathy;
* 16.Presence of ascites detectable on physical examination, ascites causing clinical symptoms, or ascites requiring special management during screening. Uncontrolled pleural effusion or pericardial effusion during screening;
* 17.Active gastrointestinal bleeding or a documented history of gastrointestinal bleeding within 6 months before the first dose; history of gastrointestinal perforation and/or fistula, or history of gastrointestinal obstruction within 6 months before the first dose;
* 18.History of major surgery within 4 weeks before the first dose (procedures such as central venous catheterization, needle biopsy, and feeding tube placement are not considered major surgery);
* 19.History of solid organ or hematopoietic stem cell transplantation;
* 20.Past or current non-infectious pneumonia/interstitial lung disease requiring systemic glucocorticoid treatment;
* 21.Cardiac dysfunction, including:

  1. Diagnosis of long QT syndrome, or QTcF (corrected QT interval using Fridericia's formula) ≥ 450 ms in males and ≥ 470 ms in females during screening (only one ECG recheck is permitted during screening, with the result of the last ECG in the screening period taken as final);
  2. High-grade atrioventricular block;
  3. Malignant arrhythmia poorly controlled by medication;
  4. History of chronic heart failure with NYHA (New York Heart Association) functional class ≥ 3;
  5. Severe valvular heart regurgitation or stenosis requiring treatment;
  6. Acute coronary syndrome or severe myocardial disease (including primary cardiomyopathy and other severe myocardial diseases assessed by the investigator) within 6 months prior to screening; severe pericardial disease (including acute pericarditis, constrictive pericarditis and other severe pericardial diseases assessed by the investigator) within 6 months prior to screening;
  7. Left ventricular ejection fraction (LVEF) < 50% as indicated by echocardiography;
* 22.History of severe neurological or psychiatric disorders (including epilepsy or dementia) that affect trial compliance;
* 23.Limb vascular thrombosis with potential severe consequences detected by ultrasound during screening; or history of thromboembolic events within 12 months prior to enrollment;
* 24.Participants with severe bleeding tendency, or history of major bleeding events within the past 6 months (e.g., previous intracranial hemorrhage, gastrointestinal bleeding, or purpura);
* 25.Urinary protein ≥ 1 g/24 h. Participants with proteinuria > 1+ on urinalysis will undergo 24-hour urine collection for quantitative assessment of proteinuria;
* 26.Other conditions deemed by the investigator to potentially increase participant risk or interfere with trial results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2025-12-23 (Estimated); Primary Completion 2028-06-26 (Estimated); Study Completion 2029-02-03 (Estimated)

PRIMARY OUTCOMES:
Phase Ib-DLT | 3years
  Incidence of Dose-Limiting Toxicity
Phase Ib- AE | 3years
  Adverse Event
Phase II- ORR | 3years
  Overall Response Rate

SECONDARY OUTCOMES:
Phase Ib- ORR | 3years
  Overall Response Rate
Phase Ib- DCR | 3years
  Disease Control Rate
Phase Ib- DoR | 3years
  Duration of Response
Phase Ib- TTR | 3years
  Time to Response
Phase Ib-PFS | 3years
  Progression-Free Survival
Phase Ib- OS | 3years
  Overall Survival
Phase Ib-PK：plasma concentration of Paclitaxel, DOTAP, Enlonstobart | 3years
  Pharmacokinetics：plasma concentration of Paclitaxel, DOTAP, Enlonstobart
Phase Ib- ADA | 3years
  Anti-Drug Antibodies
Phase Ib- Nab | 3years
  Neutralizing Anti-Drug Antibodies
Phase II- PFS | 3years
  Progression-Free Survival
Phase II- DCR | 3years
  Disease Control Rate
Phase II- DoR | 3years
  Duration of Response
Phase II- TTR | 3years
  Time to Response
Phase II-ORR | 3years
  Overall Response Rate
Phase II- OS | 3years
  Overall Survival
Phase II- TEAE | 3years
  Treatment-Emergent Adverse Event
Phase II- SAE | 3years
  Serious Adverse Event
Phase II-PK：plasma concentration of Paclitaxel, DOTAP, Enlonstobart | 3years
  Pharmacokinetics：plasma concentration of Paclitaxel, DOTAP, Enlonstobart
Phase II- ADA | 3years
  Anti-Drug Antibodies
Phase II- Nab | 3years
  Neutralizing Anti-Drug Antibodies